# PHREG - Pediatric Hypertension Registry Protocol 01/03/19 PI Andrew M. South, MD, MS Study Coordinator Lauren Vannoy

#### Background

Pediatric hypertension is increasingly common and is a precursor for adult cardiovascular and renal disease. But even during childhood, hypertension is associated with significant morbidity, including cognitive impairment and organ damage. However, the cause of pediatric hypertension, the response to treatment, and the mechanisms behind organ damage are incompletely understood. Due to these limitations, there are no first-line medications, and treatment is often inadequate. An improved comprehension of the course of pediatric hypertension could enhance clinical care. The goal of this proposal is to create a registry of patients with pediatric hypertension to better enable research into this important disease. This patient registry will enhance our ability to quickly collect and analyze data for research studies.

### Study Design

Inclusion and Exclusion CriteriaWe will include all subjects evaluated at the Brenner Children's Hospital Pediatric Nephrology clinic since January 1<sup>st</sup>, 2013 with a diagnosis of hypertension 1) confirmed with three separate blood pressure measurements ≥90<sup>th</sup> %ile for age, sex, and height, or ≥120/80 or 2) by ambulatory blood pressure monitoring with blood pressure mean <95<sup>th</sup> %ile, blood pressure load <25%, or nocturnal dipping <10%. We will also include patients from Brenner's Enhanced Care Team database using the same criteria. We will exclude patients whose initial evaluation occurred on or after their 18<sup>th</sup> birthday. An additional site, Emory University Pediatric Nephrology will be using the same criteria to enroll subjects.

## Retrospective Assessment

Brenner Children's Hospital Pediatric Nephrology will utilize i2b2 to identify our retrospective hypertension cohort. We will search for diagnosis codes of hypertension and related terms to retrospectively identify patients to be entered into the database. We anticipate a sample size of 500 subjects to be identified retrospectively at each site. Additional study sites may use i2b2 to identify subjects or a similar cohort at its discretion.

## Prospective Assessment

Sites will recruit from patients prospectively seen in their Pediatric Nephrology clinics with a diagnosis of hypertension. We will obtain parental consent and subject assent for all enrolled subjects. There are no study-specific assessments or visits. No patient biologic samples will be collected. We anticipate enrolling 200 subjects per year.

#### Data Collection

Clinical data will be collected from the electronic medical record, including sex, parent-reported race, height, weight, body mass index, age at diagnosis, age at each visit, and past medical and family histories. We will define overweight/obesity as a body mass index ≥85<sup>th</sup> %ile for age and sex. We will record systolic and diastolic blood pressure and results of ambulatory blood pressure monitoring. We will note antihypertensive medication type and dosage. We will record standard clinical laboratory values, including sodium, potassium, chloride, CO₂, blood urea nitrogen, creatinine, uric acid, aspartate aminotransferase, alanine aminotransferase, lipid profile, vitamin D 25-OH, Hgb A1c, renin, aldosterone, thyroid stimulating hormone, free thyroxine, urine albumin, urine protein, urine creatinine, and presence of hematuria. We will calculate glomerular filtration rate to measure renal function standardized to age, sex, and height. We will record results of echocardiograms, renal ultrasounds, abdominal ultrasounds

with elastography, and vesicoureterograms. Every subject will be assigned a study ID, and all data will be de-identified and stored securely ina RedCap database that will be shared across study sites and that can store site-specific patient data separately.

### References

- 1. The Fourth Report on the diagnosis, evaluation, and treatment of high blood pressure in children and adolescents. *Pediatrics* 2004; 114(Supplement 2):555-576
- 2. Din-Dzietham R, Liu Y, Bielo M-V, Shamsa F. High blood pressure trends in children and adolescents in national surveys, 1963 to 2002. *Circulation* 2007; 116(13):1488-1496. doi:10.1161/circulationaha.106.683243
- 3. Richey P, DiSessa T, Somes G, Alpert B, Jones D. Left ventricular geometry in children and adolescents with primary hypertension. *Am J Hypertens* 2010; 23:24-29
- 4. Assadi F. Effect of microalbuminuria lowering on regression of left ventricular hypertrophy in children and adolescents with essential hypertension. *Pediatric Cardiology* 2007; 28(1):27-33. doi:10.1007/s00246-006-1390-4
- 5. South AM, Arguelles L, Finer G, Langman C. The renin profile in predicting blood pressure response to treatment of essential hypertension in children [abstract]. Paper presented at the American Society of Pediatric Nephrology Annual Meeting, Boston, MA, April 28 May 1 2012 6. Washburn LK, Nixon PA, Russell GB, Snively BM, O'Shea TM. Preterm birth is associated with higher uric acid levels in adolescents. *J Pediatr* 2015; 167(1):76-80. doi:http://dx.doi.org/10.1016/j.jpeds.2015.03.043
- 7. Feig DI, Soletsky B, Johnson RJ. Effect of allopurinol on blood pressure of adolescents with newly diagnosed essential hypertension: a randomized trial. *JAMA : the journal of the American Medical Association* 2008; 300(8):924-932. doi:10.1001/jama.300.8.924
- 8. Mazzali M, Hughes J, Kim Y-G, et al. Elevated uric acid increases blood pressure in the rat by a novel crystal-independent mechanism. *Hypertension* 2001; 38(5):1101-1106. doi:10.1161/hy1101.092839
- 9. Kuczmarski R, Ogden C, Guo S, et al. 2000 CDC Growth Charts for the United States: methods and development. *Vital Health Stat 11* 2002; 246:1-190
- 10. Schwartz GJ, Brion LP, Spitzer A. The use of plasma creatinine concentration for estimating glomerular filtration rate in infants, children, and adolescents. *Pediatr Clin North Am* 1987; 34(3):571-590
- 11. Flynn JT, Daniels SR, Hayman LL, et al. Update: ambulatory blood pressure monitoring in children and adolescents. *A Scientific Statement From the American Heart Association* 2014; 63(5):1116-1135. doi:10.1161/hyp.00000000000000000
- 12. Khoury PR, Mitsnefes M, Daniels SR, Kimball TR. Age-specific reference intervals for indexed left ventricular mass in children. *Journal of the American Society of Echocardiography* 2009; 22(6):709-714. doi:http://dx.doi.org/10.1016/j.echo.2009.03.003
- 13. Rademacher ER, Sinaiko AR. Albuminuria in children. *Curr Opin Nephrol Hypertens* 2009; 18(3):246-251